CLINICAL TRIAL: NCT04770818
Title: Lateral Ankle Ligament Reconstruction With InternalBrace™ Augmentation: A Prospective Randomized Study
Brief Title: Lateral Ankle Ligament Reconstruction With InternalBrace™ Augmentation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Arthrex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 928
Record Dates: First submitted 2021-02-02; First posted 2021-02-25 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Lateral Ankle Instability

STUDY DESIGN:
Intervention Model Description: Subject is randomized to one of two arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Modified Brostrum procedure (Active Comparator): Lateral ankle ligament stabilization procedure utilizing two 2.4mm BioComposite SutureTaks to repair the ATFL (anterior talo-fibular ligament), CFL (calcanealfibular ligament), lateral ankle capsule and extensor retinaculum.
  Interventions: Device: Modified Brostrum procedure
- Modified Brostrum procedure with InternalBrace ligament augmentation (Active Comparator): Lateral ankle ligament stabilization procedure utilizing two 2.4mm BioComposite SutureTaks to repair the ATFL, CFL, lateral ankle capsule and extensor retinaculum with InternalBrace fixation using a 4.75mm BioComposite SwiveLock.
  Interventions: Device: Modified Brostrum procedure with Internal Brace Augmentation

INTERVENTIONS:
Device: Modified Brostrum procedure with Internal Brace Augmentation — Open, anatomic repair of the anterior talofibular and calcaneofibular ligaments for lateral ankle stability with InternalBrace augmentation.
  Arms: Modified Brostrum procedure with InternalBrace ligament augmentation
Device: Modified Brostrum procedure — Open, anatomic repair of the anterior talofibular and calcaneofibular ligaments for lateral ankle stability
  Arms: Modified Brostrum procedure

SUMMARY:
Lateral ankle ligament stabilization procedures are well described in the orthopaedic literature. Although success rates are high, the incidence of recurrent instability is well documented. In addition, with standard rehabilitation protocols, the timeline to return to sport and functional activities may be prolonged. The InternalBrace Ligament Augmentation Repair is a safe and reproducible technique using FiberTape® and BioComposite SwiveLock® as an augmentation to a Brostrom procedure. The InternalBrace Ligament Augmentation repair consists of a FiberTape bridge between two Knotless Swivelock anchors providing a protective reinforcement and allows the surgeon to repair lateral or medial ankle instability and the pain associated with it. This type of repair can be utilized in acute and chronic ankle sprains.

DETAILED DESCRIPTION:
It is hypothesized that use of InternalBrace Ligament Augmentation in addition to standard anatomic modified Brostrum repair allows for earlier return to pre-injury level compared to a standard Brostrum procedure. It is also secondarily hypothesized that intermediate and long term incidence of recurrent instability will be lower with use of internal brace augmentation of standard modified Brostrum lateral ankle ligament reconstruction.

ELIGIBILITY:
Inclusion criteria

* Subjects that consent to the study
* Ages 18 and older
* Subjects who are candidates for primary ankle instability reconstruction utilizing a standard Brostrum technique
* Able to understand, complete and sign/date the Informed Consent Form (ICF)

Exclusion criteria

* Subjects that are pregnant or planning to become pregnant within 58 weeks after surgery
* Persons with a mental or cognitive disability deemed significant enough that they would not be capable of completing the outcome measures
* Systemic laxity
* Bony correction (i.e. calcaneal osteotomy)
* Major additional tendon surgery such as tenodesis or repair of the peroneal tendon (synovectomy is allowable)
* Major arthroscopic surgery such as treatment of chondral defects, including microfracture (arthroscopic synovectomy and arthroscopically treated osteophyte resection are allowable)
* Revision surgery
* Inadequate tissue for standard Brostrum reconstruction
* Neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2016-03-10 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2023-03-10 (Estimated)

PRIMARY OUTCOMES:
Return to Work | Subject is called every 2 weeks between 6-26 weeks post-op timepoint and asked when they returned to pre-injury level.
  Subject self-assessment of time of return to pre-injury level.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | Data collected at the following time points: Pre-operative, 3 weeks, 6 weeks, 12 weeks, 26 weeks, 1 year, 2 years, 3 years, 4 years, 5 years
  The VAS is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" (0) and "worst pain (10).
Veterans Rand (VR-12) | Data collected at the following time points: Pre-operative, 6 weeks, 12 weeks, 26 weeks, 1 year, 2 years, 3 years, 4 years, 5 years
  The VR-12 is a patient-reported instrument from which physical and mental health component summary scores (Physical Component Score and Mental Component Score) are derived. The VR-12 items assess physical functioning, role limitations due to physical or mental health problems, pain, energy, mental health, social functioning, and general health. The United States population average PCS and MCS are both 50 points. The United States population standard deviation is 10 points. Therefore, each increment of 10 points above or below 50 corresponds to one standard deviation away from the population average. Change from pre-op and post-operative data collection timepoints will be assessed.
Foot and Ankle Ability Measure (FAAM) | Data collected at the following time points: Pre-operative, 6 weeks, 12 weeks, 26 weeks, 1 year, 2 years, 3 years, 4 years, 5 years
  The FAAM is a self-report measure that assesses physical function of individuals with lower leg, foot, and ankle musculoskeletal disorders. The Foot and Ankle Ability Measure is a 29-item questionnaire divided into two subscales: the 21-item Activities of Daily Living Subscale and the 8-item Sports Subscale. Each item is scored on a 5-point Likert scale (4 to 0) from 'no difficulty at all' to 'unable to do'. Item score totals, which range from 0 to 84 for the ADL subscale and 0 to 32 for the Sports subscale, were transformed to percentage scores. Higher scores represent higher levels of function for each subscale, with 100% representing no dysfunction. Change from pre-op and post-operative data collection timepoints will be assessed.
Karlsson and Peterson Scoring System | Data collected at the following time points: Pre-operative, 6 weeks, 12 weeks, 26 weeks, 1 year, 2 years, 3 years, 4 years, 5 years
  TheKarlsson and Peterson Scoring System is a self-report that assesses ankle function. It is composed of 8 questions with a low score of 0 (low function) and a high score of 100 (high function). Change from pre-op and post-operative data collection timepoints will be assessed.
Tegner Activity Score | Data collected at the following time points: Pre-operative, 6 weeks, 12 weeks and 26 weeks.
  The Tegner activity scale is a one-item score that grades activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer. Change from pre-op and post-operative data collection timepoints will be assessed.
Range Of Motion | Data collected at the following time points: Pre-operative, 6 weeks, 12 weeks, 26 weeks and 1 year.
  Range of motion of joints is measured using an instrument called a goniometer. Range of Motion will be measured using a goniometer during passive motion in a seated position. All measurements are from a neutral position. Normal values for the ankle are 0-50 degrees for plantar flexion and 0-20 degrees for dorsiflexion. For the foot, normal values are 0--35 degrees for inversion and 0-25 degrees for eversion. Change from pre-op and post-operative data collection timepoints will be assessed.
Return to Sports | Data collected at the following time points: 6 weeks, 12 weeks and 26 weeks
  Physician assessment of patient's return to sports. Yes or No response.
Stress X-ray | Data will be collected at Pre-op and 1 year.
  A comparison of change in the anterior drawer and talar tilt. These findings determine the stability of the ligaments, The anterior drawer is measured in millimeters and the talar tilt is measured in degrees.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Illinois Bone & Joint Institute, Chicago, Illinois
  - Desert Orthopaedic Center, Las Vegas, Nevada
  - Logan Regional Orthopedics, Logan, Utah

IPD SHARING:
Plan to Share IPD: No